CLINICAL TRIAL: NCT01752439
Title: Randomized Double-Blind Sham-Controlled Study of the Effects of Transcranial Direct Current Stimulation in Refractory Chronic Migraine and Medication-overuse Headache Patients
Brief Title: Effects of Transcranial Direct Current Stimulation in Refractory Chronic Migraine and Medication-overuse Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr Armando Perrotta, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr Armando Perrotta, MD, PhD, MD, PhD, Mediterranean Neurological Institute
Organization: Mediterranean Neurological Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCSCMMOH1
Record Dates: First submitted 2012-12-11; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Migraine; Medication Overuse Headache
Keywords: Chronic Migraine; Medication Overuse Headache; Refractory; transcranial direct current stimulation
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anodal transcranial direct current stimulation (Experimental): Anodal transcranial direct current stimulation
  Interventions: Device: Anodal transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Sham transcranial direct current stimulation
  Interventions: Device: Sham transcranial direct current stimulation
- Control group (No Intervention)

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation
  Other Names: Transcranial direct current stimulator HDCstim, Newronika s.r.l., Milan, Italy
  Arms: Anodal transcranial direct current stimulation
Device: Sham transcranial direct current stimulation
  Other Names: Transcranial direct current stimulator HDCstim, Newronika s.r.l., Milan, Italy
  Arms: Sham transcranial direct current stimulation

SUMMARY:
The purpose of the study is to evaluate the efficacy of the transcranial direct current stimulation of the primary motor cortex (M1) in patients affected by refractory chronic migraine (coded as 1.5.1 in the international headache classification 2nd edition, 2004) and medication-overuse headache (coded as 8.1) with migraine as primary headache.

ELIGIBILITY:
Inclusion Criteria:

* Chronic MIgraine or Medication Overuse Headache according to the diagnostic criteria set out in the 2nd edition of the International Classification of Headache Disorders refractory to treatment according to the Refractory Headache Special Interest Section of the American Headache Society (Schulman et al., 2008)

Exclusion Criteria:

* Other primary or secondary headaches.
* Any serious systemic or neurological disease or psychiatric disorder.
* Pregnancy or breastfeeding
* Previous or current use of other or similar devices for pain control
* Heart conduction and rhythm disorders
* Cranial surgery
* Other pain conditions, accordingly with current guidelines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in headache days per months | at 30, 60 and 90 days after the treatment
Change in drugs intake per months | at 30, 60 and 90 days after treatment

SECONDARY OUTCOMES:
Change in mean pain intensity score per months | at 30, 60 and 90 days after treatment